CLINICAL TRIAL: NCT07141901
Title: Improving Colorectal Cancer Screening Decisions Through Consideration of Life Expectancy
Brief Title: Life Expectancy-informed Colorectal Cancer Screening
Acronym: CRC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathryn Martinez (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Kathryn Martinez, Associate Staff, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 24-1038; R01AG086247 (NIH)
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer Control and Prevention
Keywords: life expectancy; colorectal cancer; screening; preventative; decision support tool
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): For patients with life expectancy <10 years: Active (i.e. interruptive) BPA that will fire when the clinician orders colorectal cancer screening. The BPA will advise that screening is not recommended due to <10 year life expectancy. An active alert is required to prevent the clinician from ordering a potentially inappropriate test. The BPA will contain a box with suggested language with which to express this to the patient.
  For patients with life expectancy ≥10 years: Passive alert on the Storyboard indicating that patient could benefit from screening as their predicted life expectancy is ≥10 years. A passive alert does not interfere with workflow and is available whenever it is convenient for the clinician to address it.
  Interventions: Behavioral: Decision Tool
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Decision Tool — For patients with life expectancy <10 years: Active (i.e. interruptive) BPA that will fire when the clinician orders colorectal cancer screening. The BPA will advise that screening is not recommended due to <10 year life expectancy. An active alert is required to prevent the clinician from ordering a potentially inappropriate test. The BPA will contain a box with suggested language with which to express this to the patient.
  For patients with life expectancy ≥10 years: Passive alert on the Storyboard indicating that patient could benefit from screening as their predicted life expectancy is ≥10 years. A passive alert does not interfere with workflow and is available whenever it is convenient for the clinician to address it.
  Arms: Intervention

SUMMARY:
The purpose of this study is to improve life-expectancy concordant colorectal cancer screening for adults over 75 years through design and testing of a life expectancy notification to clinicians delivered via the electronic health record.

This study has three components:

1. The investigators will develop a life expectancy prediction model using patient data from the Cleveland Clinic electronic health record (EHR) and test it against two existing life expectancy prediction models to determine which should be used in clinical care. This is an observational cohort study.
2. Concurrently with the development and testing of the life expectancy prediction model, the investigators will conduct interviews with clinicians to generate knowledge regarding the optimal way to integrate life expectancy information into decision making about colorectal cancer screening in patients over 75 years. This is a qualitative study.
3. The investigators will then conduct a cluster randomized trial of a clinical decision support-delivered life expectancy notification on life expectancy-congruent colorectal cancer screening orders by primary care clinicians.

DETAILED DESCRIPTION:
The purpose of this study is to improve life-expectancy concordant colorectal cancer screening for adults over 75 years through design and testing of a life expectancy notification to clinicians delivered via the electronic health record.

The investigators will pull patient data from the Cleveland Clinic Electronic Health Record (EHR) and use this to build and test a prediction model. The investigators will compare this model against two other existing life expectancy prediction models using these data. Once the investigators have identified the model with the best predictive ability, the investigators will test the model in the Metro Health System study population.

Concurrently with the development and testing of the life expectancy prediction model, the study team will develop the interview guide, which will be semi-structured; the investigators will use pre-defined questions based on study interest but will also allow for new topics to emerge. The investigators will invite clinicians for interviews based on their prior two-year colonoscopy ordering for patients >75 years, identifying clinicians in the top quarter and bottom quarter of colonoscopy orders compared to their peers. Akin to a "positive deviance" sampling approach, this method will capture clinician perspectives at both ends of the distribution and will provide richer information about how varied clinicians consider life expectancy in colonoscopy decision making. As the investigators want to collect diverse clinician perspectives, unique clinicians will be recruited for each phase of interviews. Interviews will last between 45 minutes and an hour take place via Microsoft Teams. Interviews will be audio recorded and transcribed verbatim. For each phase, following coding of 10 interviews, investigators will share findings with the study team and develop a preliminary coding dictionary. Subsequent interviews will be coded using this dictionary, adding additional codes as they emerge. Interviews will continue until thematic saturation is reached. Based on prior similar studies the investigators anticipate this will require 20 clinician interviews per phase.

The investigators will work with the Cleveland Clinic EHR team to implement the life expectancy algorithm and the Best practice alerts (BPA) into EHR. The BPAs will be piloted over a one-month period by 10 clinicians. During the pilot, the investigators will monitor use to ensure the BPAs are working correctly, in keeping with the 5 Rights framework. (e.g. displaying for the right patients in the right location). The investigators will conduct clinician interviews to elicit feedback on the notification, including making changes to the suggested language to support screening discontinuation for patients with <10 years life expectancy. The investigators will then modify the placement and/or the wording of the notifications and conduct another pilot. Based on experience, 1-2 pilots will be sufficient, but the investigators can conduct a third round, if needed.

The investigators will randomize the clinics 3:2, with 30 sites in the intervention arm and 20 sites in the control arm. The investigators will then turn on the Clinical Decision Support at the intervention sites, where it will fire automatically for any eligible patient. By pulling data from the EHR, the investigators will assess colonoscopy orders, and other outcomes between 1 and 365 days following the index visit.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1a: Patients must meet all the inclusion criteria listed below to be included:

  * > 75 years of age
  * Resident of Ohio
  * Had at least one Internal Medicine or Family Medicine visit at Cleveland Clinic Health System between January 1, 2007, and September 1, 2022.

Aim 1b: Clinicians must meet all the inclusion criteria listed below to be included:

* Internal Medicine or Family Medicine clinician (MD, DO, or APP) practicing at Cleveland Clinic Health System in Northeast Ohio
* Saw ≥10 study-eligible patients, defined as patients aged >75 years who were due or overdue for colorectal cancer screening, between 2024-2025
* With a colonoscopy ordering rate for patients >75 years in either the top quarter of the distribution of all eligible clinicians or bottom quarter of all eligible clinicians

Aim 2: Clinics must meet all the inclusion criteria listed below to be included:

• Internal Medicine or Family Medicine clinical site included in the Cleveland Clinic Health System in Northeast Ohio or Florida

Clinicians must meet all the inclusion criteria listed below to be included:

* Currently practicing in Internal or Family Medicine as an attending clinician
* Saw ≥10 study-eligible patients, defined as patients aged >75 years who were due or overdue for colorectal cancer screening, between 2024-2025

Patients must meet all the inclusion criteria listed below to be included:

* >75 years of age
* Have not received a colonoscopy in the prior 10 years
* Have not received a FOBT/FIT in prior year
* Had a visit in Internal Medicine or Family Medicine between January 1, 2026 and January 1, 2028

Exclusion Criteria:

* All candidates meeting any of the exclusion criteria at baseline will be excluded from study participation.

Aim 1a:

* Patients aged ≤75 years
* Patients who did not have at least one subsequent Internal or Family Medicine visit in Ohio within two years from the date of their baseline visit
* Patients being actively treated for non-skin cancer

Aim 1b:

* Clinicians who are not in the top or bottom quarter of the distribution of colonoscopy orderers for patients aged >75 years
* Trainees/residents
* Saw <10 study-eligible patients between 2024-2025

Aim 2:

* Patients aged <75 years
* Patients up to date with colorectal cancer screening (colonoscopy within 10 years or FOBT/FIT/Cologuard within the past year)

Min Age: 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Life-expectancy congruent colonoscopy ordering at the clinic level | 7 days
  The investigators will define this separately for patients with <10 years life expectancy and those with ≥10 years life expectancy. For both groups, the investigators will assess the proportion who received an order for colonoscopy versus not. The investigators hypothesize the intervention will result in more life expectancy-appropriate ordering: for those in the <10-year life expectancy group, the intervention will be associated with a lower ordering rate, while in the ≥10-year life expectancy group, the intervention will be associated with a higher ordering rate. The investigators will measure colonoscopy orders within 7 days of their index visit.

SECONDARY OUTCOMES:
ordering of fecal occult blood tests (FOBT) or fecal immunochemical testing (FIT), colonoscopies performed, colorectal cancers/advanced adenomas detected, polyps removed, cancers treated, and perforations | 10 days
  For patients who underwent colonoscopy, the investigators will assess the rate of hospitalization within 10 days, compared to hospitalizations within 10 days of the half-birthdays of patients who did not undergo colonoscopy. The investigators will assess the proportion of patients in each study arm for whom a colonoscopy was either recommended/not recommended by their clinicians who chose the opposite course of action.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Martinez, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared in compliance with institutional policies, IRB approval, and applicable laws and regulations (including the HIPAA Privacy Rule). Certain variables may be excluded based on organizational policies or legal requirements, such as data for which participant consent was not obtained or data that could potentially identify participants.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified data will be available to the research community after the later of:
  The end of the grant award, The publication of resulting manuscripts, or Institutional approval to share data.
  In accordance with Cleveland Clinic policy, the data will remain available for six years following study completion.
Access Criteria: Researchers may request data directly from the Principal Investigator at Cleveland Clinic. Each request will be reviewed individually with input from the Principal Investigator, the Law Department, and the Institutional Review Board (IRB).
  * Data may only be used for academic research purposes.
  * Use for commercial purposes or by individuals affiliated with for-profit institutions is prohibited.
  * Only qualified users will be granted access.
  * Users must:
  Accept a legal disclaimer. Refrain from attempting to identify participants. Obtain IRB approval or a determination that IRB approval is not required.
  Additional requirements may apply to ensure compliance with NIH policy, IRB requirements, HIPAA, and other applicable laws and regulations.